CLINICAL TRIAL: NCT02696018
Title: Evaluation of Diaphragmatic Displacement During Spontaneous Breathing Trials in Critically Ill Patients
Brief Title: Diaphragmatic Echography in Critically Ill patientS
Acronym: DECIS
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Dr, Università degli Studi di Ferrara
Other Study IDs: 138-2012
Record Dates: First submitted 2016-02-13; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Respiratory Failure
Keywords: Diaphragm; Ultrasound; Critically ill patients
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill patients: Ultrasonography in critically ill patients in weaning from mechanical ventilation
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Ultrasonographic assessment of the diaphragm function

SUMMARY:
Acute respiratory failure (ARF) is characterised by a discrepancy between load imposed on respiratory muscles and their capacity. Recently, diaphragmatic ultrasonography has been introduced in the clinical practice to evaluate diaphragmatic function. In particular, the investigators will focus on Diaphragmatic Displacement measured by M-mode ultrasonography. The aim of this study was to compare the diaphragmatic displacement with traditional weaning parameters in potentially ready to be extubated patients undergoing a spontaneous breathing trial (SBT).

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated since more than 24 hours
* clinical improvement of the underlying acute cause of the respiratory failure
* adequate cough reflex
* absence of excessive and/or purulent tracheobronchial secretion
* stable cardiovascular status
* stable metabolic status
* adequate pulmonary function
* adequate mentation

Exclusion Criteria:

* age <18 years
* pregnancy
* presence of thoracostomy, pneumothorax or pneumomediastinum
* presence of flail chest or rib fractures
* neuromuscular disease
* use of muscle-paralyzing agents within 48 hours before the study
* history or new detection of paralysis or paradoxical movement of a single hemi-diaphragm on diaphragm ultrasonography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients undergoing a spontaneous breathing trial
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Weaning success | within the first 48 hours after the spontaneous breathing trial
  A successful weaning attempt was registered when patients were extubated and breathed spontaneously for more than 48 hours. The reinstitution of mechanical ventilation at the end of spontaneous breathing trial, reintubation within 48 hours or non-invasive ventilation (NIV) support after extubation defined a failed weaning attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang JR, Tsai TH, Jerng JS, Yu CJ, Wu HD, Yang PC. Ultrasonographic evaluation of liver/spleen movements and extubation outcome. Chest. 2004 Jul;126(1):179-85. doi: 10.1378/chest.126.1.179. PMID 15249460
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Derived] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861